CLINICAL TRIAL: NCT01727193
Title: The Efficacy and Safety of Leflunomide or Azathioprine Therapy in Myasthenia Gravis Patients After Expand Thymectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Weibin, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-LEF
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; leflunomide
MeSH Terms: conditions — Myasthenia Gravis | interventions — Azathioprine; Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azathioprine (Active Comparator): cholinesterase inhibitors+Glucocorticoid +Azathioprine
  Interventions: Drug: Azathioprine
- Leflunomide (Active Comparator): cholinesterase inhibitors+glucocorticoid+Leflunomide
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Azathioprine — The basic therapy of each group is cholinesterase inhibitors (pyridostigmine 36mg / kg / d). Group 1 glucocorticoid + Azathioprine: Glucocorticoid (0.25mg/kg/d )plus Azathioprine at a starting dose of 50mg/d for 14 days, then increase up to 2mg/kg in 2 weeks.If no adverse events occurred , maintain the dose until 48 weeks.
  Arms: Azathioprine
Drug: Leflunomide — The basic therapy of each group is cholinesterase inhibitors (pyridostigmine 36mg / kg / d). Group 2 glucocorticoid + Leflunomide: Glucocorticoid (0.25mg/kg/d )plus Leflunomide 20mg/d for adult, 10mg/d for child. if no adverse events occurred , maintain the dose until 48 weeks.
  Arms: Leflunomide

SUMMARY:
This is a randomized controlled clinical study. The investigators screen of eligible patients, randomized divide into the following two groups: corticosteroids + azathioprine group, corticosteroids + leflunomide group. The investigators treat the enrolled patients, estimate efficacy and observed the side effects according to the requirements of program. The investigators establish a clinical database for recording patients date and statistical analysis. Evaluation of short-term and long-term efficacy of thymectomized myasthenia gravis patients in the different group prove that what kind of treatment can improve the cure rate. The investigators will evaluate the acute toxicity (gastrointestinal side effects, liver and kidney dysfunction) and long-term toxicity (immune dysfunction, gonadal suppression) when the investigators apply these therapy in the treatment of different clinical types of myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

1. 12 to 65 years；
2. Myasthenia gravis:

   1. Patients who are diagnosed as generalized or ocular myasthenia gravis
   2. have experienced extended thymectomy (including thymic hyperplasia and thymoma)， no significant complications in 6 months after operation , and does not received any immunosuppressants or glucocorticoids treatments.
   3. do not applied in plasmapheresis or immunoglobulins treatment during 3 months .
   4. women of child-bearing period do not have a plan of pregnant for at least 3 year.
   5. Written consent of the patient, after informing

Exclusion Criteria:

1. The liver , kidney or glycometabolic function is abnormal
2. Seriously complications, such as infection or symptom in central nervous system,
3. The patients who suffering from malignancy or a history of malignancy, a variety of sexually transmitted diseases and HIV infection, tuberculosis infection, and other condition which need to prohibit the use of immunosuppressive patients.
4. Be allergic to leflunomide, azathioprine
5. Pregnant or suckling period woman
6. Accompanied with mental disorders and have difficult to communication
7. Experienced myasthenia crisis in 3 months.
8. suffering from clear cardiopulmonary functional and brain abnormalities
9. Have a history of refractory hypertension or peptic ulcer .
10. One of the white blood cells, hemoglobin, and platelet count obvious abnormalities

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
the percent of achieving good response | 144 weeks
  Pharmacologic Remission (PR) was the primary efficacy endpoint observed. Record the time the patient appears from the time of medication to the time of PR, and calculate the percentage of PR patients in each arm. Criteria for PR: The patient has had no symptoms or signs of MG for at least 1 year and continues to take some form of therapy for MG. There is no weakness of any muscle on careful examination by someone skilled in the evaluation of neuromuscular disease. Isolated weakness of eyelid closure is accepted. Patients taking cholinesterase inhibitors are excluded from this category because their use suggests the presence of weakness.

SECONDARY OUTCOMES:
The changes of the disease severity and the antibody titer during the follow-up | 144 weeks
  The magnitude by which QMG or ADL scores are reduced. Total amount of steroid used during the follow-up. Level of the acetylcholine receptor antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Weibin Liu, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, SUN YAT-SEN UNIVERSITY, Guangzhou, Guangdong, China